CLINICAL TRIAL: NCT05221788
Title: Effect of Goal-directed Hemodynamic Therapy on Short-term Postoperative Complications in Patients With Extensive Burns: a Single-center Randomized Controlled Trial
Brief Title: Effect of Goal-directed Hemodynamic Therapy on Short-term Postoperative Complications in Patients With Extensive Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Red Cross Hospital (Other)
Responsible Party: Principal Investigator, Liang Bing, associate chief physician, Guangzhou Red Cross Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-079-02
Record Dates: First submitted 2022-01-10; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDHT(goal-directed hemodynamic therapy) (Experimental): Compounded sodium lactate 3 ml/kg/h was given intravenously as a basal rehydration volume before induction, and 200 ml of electrolyte solution was given after induction. If stroke volume (SV) increased >10%, 200 ml of electrolyte solution was continued until SV increased <10%. After fluid shock, if SV increases <10% but MAP <65 mmHg and/or cardiac index (CI) <2.5l/min/m2 give low-dose norepinephrine continuous pumping and/or dobutamine continuous pumping. If hypotension was accompanied by hypovolemia (defined as urine output <0.5 ml /kg/h and/or heart rate (HR) more than 20% above baseline), plasma was administered until urine output and/or heart rate returned to normal. Fluid responsiveness and hemodynamic variables were reassessed at least every 15 minutes, and more frequently in cases of hemodynamic instability.
  Interventions: Procedure: Goal-directed hemodynamic therapy
- control (No Intervention): Continuous infusion of compounded sodium lactate 5-7 ml/kg/h was allowed to receive colloidal solution, norepinephrine and dobutamine at the discretion of the anesthesiologist.

INTERVENTIONS:
Procedure: Goal-directed hemodynamic therapy — Compounded sodium lactate 3 ml/kg/h was given intravenously as a basal rehydration volume before induction, and 200 ml of electrolyte solution was given after induction. If SV increased >10%, 200 ml of electrolyte solution was continued until SV increased <10%. After fluid shock, if SV increases <10% but mean arterial pressure (MAP) <65 mmHg and/or cardiac index (CI) <2.5l/min/m2 give low-dose norepinephrine continuous pumping and/or dobutamine continuous pumping. If hypotension was accompanied by hypovolemia (defined as urine output <0.5 ml /kg/h and/or heart rate more than 20% above baseline), plasma was administered until urine output and/or HR returned to normal. Fluid responsiveness and hemodynamic variables were reassessed at least every 15 minutes, and more frequently in cases of hemodynamic instability.
  Arms: GDHT(goal-directed hemodynamic therapy)

SUMMARY:
To investigate the effect of goal-directed hemodynamic management on perfusion and short-term prognosis of patients undergoing scab grafting in early stage of extensive burns.

DETAILED DESCRIPTION:
Objective: To investigate the effect of goal-directed hemodynamic management on perfusion and short-term prognosis of patients undergoing scab grafting in early stage of extensive burns.

Methods: Ninety-five patients with extensive burns undergoing early debridement grafting were randomly divided into a standard hemodynamic management group (control group) and a goal-directed hemodynamic therapy group (GDHT group), with the control group guided by conventional parameters and the GDHT group guided by SV based on Vigileo. The primary outcome were incidence of cardiac complications, pulmonary complications, neurological disease, acute kidney injury, and pain within 7 days postoperatively. Secondary outcome included microcirculatory perfusion metrics: Lactate (lac), The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2).

ELIGIBILITY:
Inclusion Criteria:

1. the age is between 18 and 65 years old;
2. the burn area ≥ 50% total burn surface area (TBSA) or the third degree wound area ≥ 20% TBSA;
3. patients will undergo the first operation after fluid resuscitation (after the shock period). The types of operation include incision decompression, escharectomy and skin grafting, and so on.

Exclusion Criteria:

1. Severe cardiac or pulmonary disease prior to the burn injury, combined with severe internal organ damage.
2. Patients or family members refusing informed consent for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac complications | within 7 days postoperatively
  Incidence of cardiac complications within 7 days of surgery (myocardial infarction (electrocardiogram (ECG) and/or troponin T serum concentration; new-onset atrial fibrillation)
Incidence of pulmonary complications | within 7 days postoperatively
  Incidence of pulmonary complications (pneumonia, pulmonary edema, pleural effusion, oxygenation index <300)
Incidence of neurological complications | within 7 days postoperatively
  Incidence of Neurological Disorders within 7 days postoperatively (Stroke and Delirium)
Incidence of acute kidney injury | within 7 days postoperatively
  defined by acute kidney injury criteria.
postoperative pain conditions | within 7 days postoperatively
  postoperative pain

SECONDARY OUTCOMES:
Blood lacate | before operation (T1)
  an indicator related to microcirculation perfusion
Blood lacate | 1 hour into the operation (T2)
  an indicator related to microcirculation perfusion
Blood lacate | 2 hours into the operation (T3)
  an indicator related to microcirculation perfusion
Blood lactate | the end of operation (T4)
  an indicator related to microcirculation perfusion
Blood lactate | 24 hours after operation (T5)
  an indicator related to microcirculation perfusion
Blood lactate | 7 days after operation
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | before operation (T1)
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | 1 hour into the operation (T2)
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | 2 hours into the operation (T3)
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | the end of operation (T4)
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | 24 hours after operation (T5)
  an indicator related to microcirculation perfusion
The central venous-arterial carbon dioxide partial pressure difference (Pcv-aCO2) | 7 days after operation
  an indicator related to microcirculation perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Yang Cao, Study Director — Guangzhou RedCross Hospital
Locations (1):
- Guangzhou RedCross Hospital, Guanzhou, Guangdong, China